CLINICAL TRIAL: NCT01947647
Title: Transdiagnostic Psychotherapy for Veterans With Mood and Anxiety Disorders
Acronym: TBT-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-018-13S; CX000845 (Other Grant/Funding Number: VA Clinical Science Career Development Award)
Record Dates: First submitted 2013-09-11; First posted 2013-09-20 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Major Depressive Disorder; Persistent Depressive Disorder; Posttraumatic Stress Disorder; Panic Disorder; Social Phobia; Specific Phobia; Generalized Anxiety Disorder; Obsessive Compulsive Disorder
Keywords: behavior therapy; Randomized Controlled Trials; Depressive Disorder; Anxiety Disorders; comorbidity
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Panic Disorder; Phobia, Social; Phobia, Specific; Generalized Anxiety Disorder; Obsessive-Compulsive Disorder; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdiagnostic Behavior Therapy (Experimental): A new transdiagnostic CBT protocol for the depressive/anxiety disorders was developed and revised through two demonstration studies and one focus group. The resulting protocol involves several primary components, including psychoeducation on the symptoms of depression and anxiety (session 1), assessment of motivation and setup of treatment plans (session 2), exposure therapy (sessions 3-15), and relapse prevention (final session). In addition to these primary components, optional modules are included to supplement exposure therapy later in treatment to address secondary symptoms (e.g., anger, sleep, hypervigilance, drinking to cope). The goal of these modules is to allow providers to tailor treatment to specific symptoms that may be present in any single or set of diagnoses that may be reducing the effects from the primary exposure approach. Session will be weekly for 45-60 minutes with homework assignments to be completed between sessions.
  Interventions: Behavioral: Transdiagnostic Behavior Therapy
- Behavioral Activation Therapy (Active Comparator): To provide an evidence-based comparison for the transdiagnostic CBT condition, a second group of participants will receive manualized BAT. In general, BAT involves teaching patients to monitor their mood and daily activities with the goal of increasing pleasant, reinforcing activities and reducing unpleasant events. In the present study, the BAT condition will be manualized, following an existing protocol in the literature. BAT will be structurally equivalent to the transdiagnostic CBT with the same session length (45-60 minutes), frequency of sessions (weekly), duration of treatment (12-16 sessions), and amount of homework.
  Interventions: Behavioral: Behavioral Activation Therapy

INTERVENTIONS:
Behavioral: Transdiagnostic Behavior Therapy — A new transdiagnostic CBT protocol for the depressive/anxiety disorders was developed and revised through two demonstration studies and one focus group. The resulting protocol involves several primary components, including psychoeducation on the symptoms of depression and anxiety (session 1), assessment of motivation and setup of treatment plans (session 2), exposure therapy (sessions 3-15), and relapse prevention (final session). In addition to these primary components, optional modules are included to supplement exposure therapy later in treatment to address secondary symptoms (e.g., anger, sleep, hypervigilance, drinking to cope). The goal of these modules is to allow providers to tailor treatment to specific symptoms that may be present in any single or set of diagnoses that may be reducing the effects from the primary exposure approach. Session will be weekly for 45-60 minutes with homework assignments to be completed between sessions.
  Arms: Transdiagnostic Behavior Therapy
Behavioral: Behavioral Activation Therapy — To provide an evidence-based comparison for the transdiagnostic CBT condition, a second group of participants will receive manualized BAT. In general, BAT involves teaching patients to monitor their mood and daily activities with the goal of increasing pleasant, reinforcing activities and reducing unpleasant events. In the present study, the BAT condition will be manualized, following an existing protocol in the literature. BAT will be structurally equivalent to the transdiagnostic CBT with the same session length (45-60 minutes), frequency of sessions (weekly), duration of treatment (12-16 sessions), and amount of homework.
  Arms: Behavioral Activation Therapy

SUMMARY:
Cognitive behavioral therapy (CBT) is a brief, efficient, and effective psychotherapy for individuals with depressive and anxiety disorders. However, CBT is largely underutilized within Veteran Affairs Medical Centers (VAMCs) due to the cost and burden of trainings necessary to deliver the large number of CBT protocols. Transdiagnostic CBT, in contrast, is specifically designed to address numerous distinct disorders within a single protocol. This transdiagnostic approach has the potential to dramatically improve the accessibility of CBT within VAMCs and therefore improve clinical outcomes of Veterans. The proposed research seeks to evaluate the efficacy of a transdiagnostic CBT by assessing clinical outcomes and quality of life in VAMC patients with depressive and anxiety disorders throughout the course of treatment and in comparison to an existing evidence-based psychotherapy, behavioral activation treatment.

DETAILED DESCRIPTION:
Objective To evaluate the transdiagnostic CBT in a randomized clinical trial (RCT) of VAMC patients with depressive/anxiety disorders by investigating its preliminary efficacy in reducing symptomatology, comorbidity, and improving quality of life compared to behavioral activation therapy (BAT) (psychotherapy control condition). Patient satisfaction and predictors of feasibility (attendance and dropout) also will be assessed.

Recruitment Strategy VAMC patients will be recruited through the Primary Care - Mental Health Integration program and CBT Clinic at the Ralph H. Johnson (RHJ) VAMC. Within these programs, all VAMC patients reporting symptoms of depression and anxiety meet with a mental health staff member to complete a diagnostic interview and self-report measures as part of their standard clinical practices. If VAMC patients endorse symptoms consistent with a depressive/anxiety disorder, the patient's interest in participating in research will be assessed and, if agreeable to research, patients will be put in contact with research staff (same day meeting and/or follow-up phone to schedule research assessment). A research assessment will be completed with the project staff to first complete consent documentation and then assess inclusion/exclusion criteria (with a targeted sample of 96 VAMC patients; > 72 completers), including a semi-structured clinical interview and self-report questionnaires focused on the psychiatric symptoms and quality of life. Participants who meet diagnostic criteria for the targeted disorders will be randomized into a study condition, and will be assigned to a project therapist. Because most VAMC patients who meet study criteria likely will present with multiple depressive/anxiety disorders, principal diagnosis, or the most impairing of the diagnosable disorders, will be used to select patients for participation. To balance diagnoses across the two conditions, a stratified random assignment based on principal diagnosis will be used for the most common principal diagnoses (MDD, PTSD, and PD).

Procedures Eligible VAMC patients will be randomized into one of two treatment conditions: transdiagnostic CBT or BAT. Both treatment conditions will include 12-16 weekly 50-minute individual psychotherapy sessions. The total number of sessions will vary slightly depending on participant needs and progress during therapy, as is common in most CBT approaches to psychotherapy (and will serve as a covariate in the outcome analyses). The general format of sessions will involve: 1) brief check-in; 2) review of materials from previous sessions; 3) review of homework assignments; 4) overview of new materials and in-session exercises; and 5) assignment of homework for next session. Attendance and homework completion will be recorded.

Randomization Procedures Participants will be randomly assigned (1:1) to one of the two study arms (n = 59 per arm) using a permuted block randomization procedure. Randomization will be stratified by principal diagnostic group and block size will be varied to minimize the likelihood of unmasking. After determining eligibility and completing consent and baseline assessment materials, enrolled participants will be assigned to treatment groups by the Project Research Assistant using a computer generated randomization scheme. Once a participant is randomized and attends the first session, they will be included in the intent-to-treat analysis. Randomization will occur at the participant level.

Transdiagnostic CBT Treatment Condition As noted above in the Preliminary Studies section, a transdiagnostic CBT protocol was developed and revised through two demonstration studies and one focus group. The resulting protocol involves several primary components, including psychoeducation on the symptoms of depression and anxiety (session 1), assessment of motivation and setup of treatment plans (session 2), exposure therapy (sessions 3-15), and relapse prevention (final session). In addition to these primary components, optional modules are included to supplement exposure therapy later in treatment to address secondary symptoms (e.g., anger, sleep, hypervigilance, drinking to cope). The goal of these modules is to allow providers to tailor treatment to specific symptoms that may be present in any single or set of diagnoses that may be reducing the effects from the primary exposure approach. Session will be weekly for 45-60 minutes with homework assignments to be completed between sessions.

BAT Control Condition To provide an evidence-based comparison for the transdiagnostic CBT condition, a second group of participants will receive manualized BAT. BAT is based on early behavioral models that suggest that decreases in positively reinforcing healthy behaviors are associated with the development of negative affect. In general, BAT involves teaching patients to monitor their mood and daily activities with the goal of increasing pleasant, reinforcing activities and reducing unpleasant events. BA is a brief treatment, can be administered in either individual or group formats, and has demonstrated reliable effectiveness across a wide range of university, community, civilian and Veteran clinical samples with depression. BAT also has been shown to be effective in the treatment of PTSD and other related depressive/anxiety disorders in Veterans. In the present study, the BAT condition will be manualized, following an existing protocol in the literature. BAT will be structurally equivalent to the transdiagnostic CBT with the same session length (45-60 minutes), frequency of sessions (weekly), duration of treatment (12-16 sessions), and amount of homework.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria involve:

* participants must be clearly competent to provide informed consent for research participation;
* participants must meet DSM diagnostic criteria for a principal diagnosis of a depressive/anxiety disorder (Panic Disorder, PTSD, Social Anxiety Disorder, Obsessive-Compulsive Disorder (OCD), Generalized Anxiety Disorder (GAD), specific phobia, major depressive disorder, or persistent depressive disorder); and
* participants must be 18 - 80 years old.

Exclusion Criteria:

Exclusion criteria involve:

* recent history (< 2 months) of psychiatric hospitalization or a suicide attempt as documented in their medical record,
* current diagnosis of substance dependence or abuse on the structured clinical interview,
* acute, severe illness or medical condition that likely will require hospitalization and/or otherwise interfere with study procedures as documented in their medical record (e.g., active chemotherapy/radiation treatment for cancer, kidney dialysis, oxygen therapy for chronic obstructive pulmonary disease),
* recent start of new psychiatric medication (< 4 weeks),
* diagnosis of traumatic brain injury (TBI) in their medical record and/or endorsement of screener questionnaire regarding the symptoms of TBI modified from the Post-Deployment Health Assessment employed by the Department of Defense, or
* diagnosis of schizophrenia, psychotic symptoms, personality disorder, and/or bipolar disorder. VAMC patients excluded due to these factors will be reconsidered for participation once the condition related to their exclusion is resolved or stabilized. Together, these inclusion/exclusion criteria should allow the vast majority of interested VAMC patients with depressive/anxiety disorders to be eligible to participate. Ineligible VAMC patients will be referred for non-study-related treatments within mental health at the RHJ VAMC.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Gros, PhD MA BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coyne AE, Gros DF. Comorbidity as a moderator of the differential efficacy of transdiagnostic behavior therapy and behavioral activation for affective disorders. Psychother Res. 2022 Sep;32(7):886-897. doi: 10.1080/10503307.2021.2022236. Epub 2022 Jan 7. PMID 34996343
- [Derived] Shapiro MO, Gros DF. Acceptability of a transdiagnostic behavior therapy in veterans with affective disorders. Psychol Serv. 2021 Nov;18(4):643-650. doi: 10.1037/ser0000490. Epub 2020 Jul 16. PMID 32673037
- [Derived] Gros DF, Oglesby ME, Wray JM. An Open Trial of Behavioral Activation in Veterans With Major Depressive Disorder or Posttraumatic Stress Disorder in Primary Care. Prim Care Companion CNS Disord. 2019 Oct 3;21(5):19m02468. doi: 10.4088/PCC.19m02468. PMID 31600432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 105 participants were consented and completed the intake procedures. However, of the 105 total participants, 12 participants did not met eligibility for the treatment trial and were not randomized to a treatment condition.
Groups:
- Transdiagnostic Behavior Therapy: Transdiagnostic Behavior Therapy, a 12-week transdiagnostic psychotherapy for symptoms of depression and anxiety.
- Behavioral Activation: Behavioral Activation, a 12-week psychotherapy for depressive symptoms
Period: Treatment Phase
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
Started | 46 | 47
Completed | 29 | 21
Not Completed | 17 | 26
Period: 6-month Followup Phase
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
Started | 29 | 21
Completed | 20 | 13
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Transdiagnostic Behavior Therapy: Transdiagnostic Behavior Therapy is a 12-week transdiagnostic psychotherapy for symptoms of depression and anxiety
- Behavioral Activation: Behavioral Activation is a 12-week psychotherapy for symptoms of depression
- Total: Total of all reporting groups
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.46 (11.55) | 42.60 (12.91) | 43.02 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 37 | 34 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 16 | 41
  White | 17 | 27 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
DASS-Depression [Mean (Standard Deviation); unit: units on a scale] — The DASS-Depression (Lovibond and Lovibond, 1995) is a 7-item measure designed to assess dysphoric mood. Items are rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale (range 0-21). Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance. Support for the factor structure, convergent and discriminant validity, and internal consistency of the DASS has been found in community (Lovibond and Lovibond, 1995).
  units on a scale | 10.30 (6.11) | 10.54 (4.71) | 10.42 (5.41)
DASS-Anxiety [Mean (Standard Deviation); unit: units on a scale] — The DASS-Anxiety (Lovibond and Lovibond, 1995) is a 7-item measure designed to assess symptoms of fear and autonomic arousal. Items are rated on a 4-point scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale (range 0-21). Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance. Support for the factor structure, convergent and discriminant validity, and internal consistency has been found in community (Lovibond and Lovibond, 1995).
  units on a scale | 8.19 (5.95) | 6.57 (4.59) | 7.37 (5.34)
DASS-Stress [Mean (Standard Deviation); unit: units on a scale] — The DASS-Stress (Lovibond and Lovibond, 1995) is a 7-item measure designed to assess symptoms of tension and agitation. Items are rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale (range 0-21). Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance. Support for the factor structure, convergent and discriminant validity, and internal consistency has been found in community (Lovibond and Lovibond, 1995).
  units on a scale | 11.27 (5.27) | 10.41 (5.03) | 10.84 (5.14)
STICSA-Cognitive [Mean (Standard Deviation); unit: units on a scale] — The STICSA-Cognitive (Ree et al., 2008) is a 11-item measure designed to assess trait cognitive anxiety. Items are rated on a 4-point scale, ranging from 1 (not at all) to 4 (very much so), with a total score range of 11-44. Higher scores are indicative of greater symptom severity, with scores above 23 considered of clinical significance. The cognitive scale have been supported by factor analysis and has been found to have high internal consistency (alphas > .87; Gros et al., 2007; 2010).
  units on a scale | 25.62 (7.58) | 23.56 (5.95) | 24.57 (6.84)
STICSA-Somatic [Mean (Standard Deviation); unit: units on a scale] — The STICSA-Somatic (Ree et al., 2008) is a 10-item measure designed to assess trait somatic anxiety. Items are rated on a 4-point scale, ranging from 1 (not at all) to 4 (very much so), with a total score range of 10-40. Higher scores indicative of greater symptom severity, with scores above 18 considered of clinical significance. The somatic scale have been supported by factor analysis and has been found to have high internal consistency (alphas > .87; Gros et al., 2007; 2010).
  units on a scale | 21.05 (7.20) | 19.18 (5.55) | 20.09 (6.44)
IIRS [Mean (Standard Deviation); unit: units on a scale] — The IIRS (Devin et al., 1983) is a 13-item scale that assesses the extent to which a disease interferes with important domains of life. Each item is rated on a 7-point Likert scale, ranging from 1 (not very much) to 7 (very much), with a total score range of 13-91. Although norms are not available for all diagnoses given the transdiagnostic nature of the IIRS, higher scores are indicative of greater impairment. The IIRS has strong psychometric properties in the previous literature in participants with physical and/or emotional health concerns (Devins et al., 2001; Devins, 2010).
  units on a scale | 51.92 (17.55) | 52.47 (16.64) | 52.19 (17.00)

OUTCOME MEASURES:

1. Primary Outcome: DASS-Depression
Description: The DASS-Depression (Lovibond and Lovibond, 1995) is a 7-item measure designed to assess dysphoric mood. Items are rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale (range 0-21). Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance. Support for the factor structure, convergent and discriminant validity, and internal consistency of the DASS has been found in community (Lovibond and Lovibond, 1995).
Time Frame: baseline, immediate post-treatment (after session 12 complete), 6-month follow-up (after session 12 complete)
Population: 43 participants dropped out of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
Number analyzed (Participants) | 29 | 21
score on a scale
  post-treatment | 3.93 (4.83) | 5.91 (4.95)
  follow-up: number analyzed (Participants) | 20 | 13
  follow-up | 4.51 (5.10) | 6.01 (5.36)

2. Primary Outcome: DASS-Anxiety
Description: The DASS-Anxiety (Lovibond and Lovibond, 1995) is a 7-item measure designed to assess symptoms of fear and autonomic arousal. Items are rated on a 4-point scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale (range 0-21). Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance. Support for the factor structure, convergent and discriminant validity, and internal consistency has been found in community (Lovibond and Lovibond, 1995).
Time Frame: baseline, immediate post-treatment (after session 12 complete), 6-month follow-up (after session 12 complete)
Population: 43 participants dropped out of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
Number analyzed (Participants) | 29 | 21
score on a scale
  post-treatment | 4.05 (4.61) | 3.86 (3.73)
  follow-up: number analyzed (Participants) | 20 | 13
  follow-up | 4.14 (4.22) | 4.15 (2.82)

3. Primary Outcome: DASS-Stress
Description: The DASS-Stress (Lovibond and Lovibond, 1995) is a 7-item measure designed to assess symptoms of tension and agitation. Items are rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), and summed to compute the total scale (range 0-21). Higher scores are indicative of greater symptom severity, with scores greater than 10 typically considered of clinical significance. Support for the factor structure, convergent and discriminant validity, and internal consistency has been found in community (Lovibond and Lovibond, 1995).
Time Frame: baseline, immediate post-treatment (after session 12 complete), 6-month follow-up (after session 12 complete)
Population: 43 participants dropped out of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
Number analyzed (Participants) | 29 | 21
score on a scale
  post-treatment | 5.94 (5.26) | 5.00 (4.25)
  follow-up: number analyzed (Participants) | 20 | 13
  follow-up | 6.29 (5.82) | 5.93 (4.09)

4. Primary Outcome: STICSA-Cognitive
Description: The STICSA-Cognitive (Ree et al., 2008) is a 11-item measure designed to assess trait cognitive anxiety. Items are rated on a 4-point scale, ranging from 1 (not at all) to 4 (very much so), with a total score range of 11-44. Higher scores are indicative of greater symptom severity, with scores above 23 considered of clinical significance. The cognitive scale have been supported by factor analysis and has been found to have high internal consistency (alphas > .87; Gros et al., 2007; 2010).
Time Frame: baseline, immediate post-treatment (after session 12 complete), 6-month follow-up (after session 12 complete)
Population: 43 participants dropped out of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
Number analyzed (Participants) | 29 | 21
score on a scale
  post-treatment | 18.10 (8.12) | 16.90 (5.26)
  follow-up: number analyzed (Participants) | 20 | 13
  follow-up | 18.05 (8.59) | 17.85 (6.20)

5. Primary Outcome: STICSA-Somatic
Description: The STICSA-Somatic (Ree et al., 2008) is a 10-item measure designed to assess trait somatic anxiety. Items are rated on a 4-point scale, ranging from 1 (not at all) to 4 (very much so), with a total score range of 10-40. Higher scores indicative of greater symptom severity, with scores above 18 considered of clinical significance. The somatic scale have been supported by factor analysis and has been found to have high internal consistency (alphas > .87; Gros et al., 2007; 2010).
Time Frame: baseline, immediate post-treatment (after session 12 complete), 6-month follow-up (after session 12 complete)
Population: 43 participants dropped out of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
Number analyzed (Participants) | 29 | 21
score on a scale
  post-treatment | 16.57 (6.90) | 16 (4.59)
  follow-up: number analyzed (Participants) | 20 | 13
  follow-up | 16.81 (5.61) | 16.96 (4.17)

6. Primary Outcome: IIRS
Description: The IIRS (Devin et al., 1983) is a 13-item scale that assesses the extent to which a disease interferes with important domains of life. Each item is rated on a 7-point Likert scale, ranging from 1 (not very much) to 7 (very much), with a total score range of 13-91. Although norms are not available for all diagnoses given the transdiagnostic nature of the IIRS, higher scores are indicative of greater impairment. The IIRS has strong psychometric properties in the previous literature in participants with physical and/or emotional health concerns (Devins et al., 2001; Devins, 2010).
Time Frame: baseline, immediate post-treatment (after session 12 complete), 6-month follow-up (after session 12 complete)
Population: Patient assigned to psychotherapy triage appointment within the MHC CBT Clinic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
Number analyzed (Participants) | 29 | 21
score on a scale
  post-treatment | 33.13 (21.31) | 33.84 (18.08)
  follow-up: number analyzed (Participants) | 20 | 13
  follow-up | 32.85 (20.41) | 29.77 (11.50)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for approximately 9-months per participants. More specifically, adverse events were monitored from baseline (week 0) through the course of the 12-session weekly treatment and until the 6-month followup assessment was completed (6-months following completion of session 12).
Arm/Group | Transdiagnostic Behavior Therapy | Behavioral Activation
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47

LIMITATIONS AND CAVEATS:
higher than expected dropout rates

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT01947647/Prot_SAP_000.pdf